CLINICAL TRIAL: NCT01466023
Title: The Reduced Thyroid Function of the Premature Newborn: Relation With Molecular Changes in the Placenta and Maternal Thyroid Hormone Status and Neurodevelopmental Implications
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S53423
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2011-07

CONDITIONS: Thyroid Metabolism
Keywords: thyroid metabolism during pregnancy; impact on neonate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Placenta and blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Transient hypothyroxinemia of prematurity (THOP) is a typical entity of the preterm infant, affecting the majority of preterm infants, born less than 30 weeks of gestational age. It is defined as a temporary postnatal reduction from cord values in serum levels of T4 and FT4, but with normal thyroid-stimulating hormone (TSH) levels.The etiology of THOP is complex and multifactorial. Loss of maternal T4, limited postnatal thermogenesis, hypothalamic-pituitary immaturity, limited thyroid gland reserve, persistent fetal thyroid hormone metabolism and predisposition to nonthyroidal illness syndrome are several factors that contribute in less or more intensity to THOP.The association between THOP and poor neurodevelopmental outcome is well established and several therapeutic clinical trials have been set up. However, there is currently no evidence for prophylactic or therapeutic supplementation with thyroxine (T4) for premature infants with THOP. One study of van Wassenaer et al. showed a beneficial effect of treatment of THOP in a subgroup of preterm infants with gestational age less than 28 weeks, but a reverse effect in the group with a gestational age of 29 weeks. This is an illustration of the limited comprehension of the pathophysiology of THOP.

Although studies about THOP usually involves the preterm infants born at 33 weeks or earlier, one study of Paul et al. showed a decreased thyroid function in late preterm and term infants with respiratory distress syndrome as function of severity of illness. Unpublished data of our center showed also the presence of THOP, although less frequent, in the group of late preterm infants. Other data about this group of preterm infants are scarce.

During the first half of pregnancy, the fetus is completely dependent of maternal thyroid hormone supply and the fetal thyroid gland starts thyroid hormone secretion from about 17-19 weeks of gestational age. Conditions of maternal (sub)clinical hypothyroidism are associated with complications like hypertension, preterm birth, low birth weight, placental abruption, and fetal death. One can wonder if there are compensating mechanisms in the placenta, providing the fetus with sufficient thyroid hormone in cases of compromised thyroid supply. One study showed that total placenta deiodinase type 3 (D3) activity in pregnancies with severely hypothyroid fetuses was not significantly lower than in euthyroid controls. Two studies showed increased monocarboxylate transporter 8 (MCT8) and decreased MCT10 expression within placentae of pregnancies complicated by IUGR. As far as we know, nothing is known about possible compensating effects in placentae of mothers with subclinical hypothyroidism and the possible influence on the development of THOP.

Maternal subclinical hypothyroidism during pregnancy is a predisposition for the development of overt hypothyroidism. The influence of maternal thyroid antibodies during pregnancy towards thyroid hormone function of the fetus and consequently neurodevelopmental outcome is still not clear. One single study of Negro et al. showed that euthyroid pregnant women who are positive for thyroid peroxidase antibodies (TPOAb) develop impaired thyroid function, which is associated with an increased risk of miscarriage and premature deliveries. They also showed that substitutive treatment with levothyroxine (LT4) is able to lower the chance of miscarriage and premature delivery.A study of Pop et al. concluded that children of pregnant women who had elevated titers of TPO-Ab but normal thyroid function are at risk for impaired development.Nothing is known about the possible influence of maternal thyroid antibodies towards the development of THOP, although a theoretical link is possible.

The investigators want to investigate whether there are compensatory mechanisms in placentas of premature born infants and whether the maternal thyroid hormone condition is a prediction of the development of THOP in the premature infant. The investigators want to investigate the differences between several groups of preterm infants: 24-28 weeks, 28-32 weeks and 32-36 weeks. The further aim of this study is to investigate the impact of maternal thyroid hormone condition during pregnancy on neurodevelopmental outcome of the neonate.

In Belgium, 8% of the newborns are born preterm. There are about 2000 deliveries each year in the University Hospitals Leuven. Between 2 and 5% of all pregnant women are considered to have subclinical hypothyroidism and preterm birth is almost 2-fold higher in women with subclinical hypothyroidism.The incidence of THOP is 30 %. We performed a statistical power calculation with a confidence level of 95%. Given the above data and with the assumption that 50% of the premature babies born to a hypothyroid mothers will develop THOP, we need to include 320 patients who give premature birth to obtain a statistical power of 80%. Therefore, the inclusion time will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* at risk of preterm delivery

Exclusion Criteria:

* known congenital abnormality

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women in a tertiairy hospital
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium